CLINICAL TRIAL: NCT06460454
Title: PROnostic Interest of 18F-FDG PET/CT in Patients With Metastatic Castration-resistant Prostate Cancer (mCPRC) Progressing on Chemotherapy, Treated With 177 Lu-PSMA (PROFLu)D7 (± 1 Day)
Brief Title: PROnostic Interest of 18F-FDG PET/CT in Patients With Metastatic Castration-resistant Prostate Cancer (mCPRC) Progressing
Acronym: PROFLu
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, BOURSIER Caroline, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2024PI101
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
Keywords: nuclear medicine; prostate cancer; PET scan
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated with 177Lu-PSMA for castration-resistant prostate cancer: Patients treated with 177Lu-PSMA for castration-resistant prostate cancer and who benefited from 68Ga-PSMA and 18FDG PET scans as part of the initial workup and treatment follow-up.
  Interventions: Device: PET scan of 18F-FDG

INTERVENTIONS:
Device: PET scan of 18F-FDG — VEREOS PET scanner. Philips VEREOS digital PET-CT scanners are installed in the nuclear medicine department.

SUMMARY:
The aim of this retrospective study was to assess the prognostic value of parameters extracted from 18FDG PET/CT and 68Ga-PSMA PET in the initial workup and follow-up of patients treated with 177Lu-PSMA in mCRPC.

DETAILED DESCRIPTION:
Prostate-specific membrane antigen (PSMA) is expressed in most metastatic castration-resistant prostate cancer (mCRPC) cells. In response to this finding, a vectorized internal radiotherapy (VIR) therapy was developed, lutetium 177-labeled PSMA, 177Lu-PSMA. Clinical trials have demonstrated its efficacy in men with metastatic castration-resistant prostate cancer . The number of patients treated in nuclear medicine departments has increased considerably in recent years, notably with the Food and Drug Administration's (FDA) and the European Medicines Agency's (EMA) approval of this treatment (177Lu-PSMA-617, Pluvicto®) in the setting of progressive mCRPC after at least one line of 2nd-generation hormone therapy and one line of taxane chemotherapy.

Patients eligible for treatment benefit from pre-therapy 68Ga-PSMA positron emission tomography (PET/CT) to assess PSMA expression by cancer cells, but 18FDG PET/CT, although mentioned in the EANM guidelines, is not routinely performed. For treatment follow-up of prostate cancer patients, the PCWG3 (prostate cancer working group 3) currently recommends conventional imaging (CT scan and bone scan) (4) and makes no mention of metabolic imaging, even though some lesions are not detectable with conventional imaging. In addition, one study reported that a high metabolic volume 18FDG PET/CT scan as part of the pre-therapy work-up for mCRPC prior to the introduction of 177Lu-PSMA or Cabazitaxel therapy was associated with a poorer response to treatment.

The aim of this retrospective study was to assess the prognostic value of parameters extracted from 18FDG PET/CT and 68Ga-PSMA PET in the initial work-up and follow-up of patients treated with 177Lu-PSMA in mCRPC.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with 177Lu-PSMA for castration-resistant prostate cancer at Nancy University Hospital
* Patients with 68Ga-PSMA and 18FDG PET scans as part of the initial workup and treatment follow-up

Exclusion Criteria:

* Patients who did not give their consent to use their data retrospectively

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients treated with 177Lu-PSMA for castration-resistant prostate cancer at the CHRU de Nancy and who benefited from 68Ga-PSMA and 18FDG PET scans as part of the initial workup and treatment follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of 18FDG PET metabolic volume | 1 year
  Diagnostic accuracy of 18FDG PET metabolic volume in predicting 1-year overall survival.

SECONDARY OUTCOMES:
Diagnostic accuracy of 18FDG PET tumor parameter (SUVmax) | 1 year
  Diagnostic accuracy of 18FDG PET tumor parameter (SUVmax) in predicting 1-year overall survival.
Diagnostic accuracy of 18FDG PET tumor parameters (SUVmean) | 1 year
  Diagnostic accuracy of 18FDG PET tumor parameters (SUVmean), in predicting 1-year overall survival.
Diagnostic accuracy of 18FDG PET tumor parameters (FDG/PSMA mismatch) | 1 year
  Diagnostic accuracy of 18FDG PET tumor parameters (FDG/PSMA mismatch) in predicting 1-year overall survival.

CONTACTS AND LOCATIONS:
Locations (1):
- Nuclear medicine Department CHRU de NANCY, Vandœuvre-lès-Nancy, France